CLINICAL TRIAL: NCT01765595
Title: Clinical and Economic Impact of an Electronic Medical Record Interfaced Decision Support System for Minimizing Severe Drug-Drug Interactions
Acronym: DDI+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leumit Health Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LHS012013
Record Dates: First submitted 2013-01-09; First posted 2013-01-10 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Healthcare
Keywords: health care expenditure; drug drug interactions; electronic decision support systems; Potential reduction

ARMS (2):
- DDI+ (Experimental): DDI+ Incorporated in routine ambulatory practice
  Interventions: Other: DDI+
- Control (No Intervention): Standard care

INTERVENTIONS:
Other: DDI+
  Arms: DDI+

SUMMARY:
Leumit Health Services, an health maintenance organization operating in Israel, will incorporate a web-based, decision support system for handling drug-drug interactions and drug information, termed DDI+. the investigators hypothesize that implementing such a system will reduce health-care expenditures (e.g., hospital admissions, referrals to ERs, Imaging procedures).

ELIGIBILITY:
Inclusion Criteria:

* Number of chronic concomitant drugs ≥5

Exclusion Criteria:

* Patients diagnosed with HIV/AIDS, and/or viral hepatitis B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 715 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Hospital Admissions | up to 12 months post initiation

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Weizman, MD, Principal Investigator — Tel Aviv University
Locations (1):
- Leumit Health Services, Tel Aviv, Israel